CLINICAL TRIAL: NCT01343082
Title: A Long-term Open-label Study of DE-111 Ophthalmic Solution in Patients With Open Angle Glaucoma or Ocular Hypertension -Phase 3-
Brief Title: DE-111 Ophthalmic Solution in Patients With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01111006
Record Dates: First submitted 2011-04-24; First posted 2011-04-27 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Open Angle Glaucoma or Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

ARMS (1):
- 1 (Experimental): DE-111 ophthalmic solution
  Interventions: Drug: DE-111 ophthalmic solution

INTERVENTIONS:
Drug: DE-111 ophthalmic solution

SUMMARY:
Safety and IOP (intraocular pressure) lowering effect of DE-111 ophthalmic solution will be evaluated in open-angle glaucoma or ocular hypertension patients, in an open-label, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open angle glaucoma or ocular hypertension
* Provided signed, written informed consent
* 20 years of age and older
* If a subject is a female of childbearing potential, she must utilize reliable contraceptive throughout the study, and must have a negative urine pregnancy test prior to enrollment into this study

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy, or females of childbearing potential who are not using a reliable method of contraception.
* Presence of any abnormality or significant illness that could be expected to interfere with the study.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The run-in period of 4 weeks. Switched to DE-111 ophthalmic solution from Tafluprost ophthalmic solution 0.0015%, Timolol ophthalmic solution 0.5%, or concomitant Tafluprost ophthalmic solution 0.0015% plus Timolol ophthalmic solution 0.5% . Treatment period: 52 weeks .
Groups:
- Allocated to Tafluprost: Switched to DE-111 ophthalmic solution (one drop at a time, once daily, bilateral topical instillation) from Tafluprost ophthalmic solution 0.0015% (one drop at a time, once daily, bilateral topical instillation) .
- Allocated to Timolol: Switched to DE-111 ophthalmic solution (one drop at a time, once daily, bilateral topical instillation) from Timolol ophthalmic solution 0.5% (one drop at a time, BID, bilateral topical instillation).
- Allocated to Tafluprost + Timolol: Switched to DE-111 ophthalmic solution (one drop at a time, once daily, bilateral topical instillation) from concomitant Tafluprost ophthalmic solution 0.0015% plus Timolol ophthalmic solution 0.5%.
Period: The run-in Period
Arm/Group | Allocated to Tafluprost | Allocated to Timolol | Allocated to Tafluprost + Timolol
Started | 51 | 49 | 48
Completed | 48 | 45 | 43
Not Completed | 3 | 4 | 5
Not completed — Not meeting criteria | 3 | 4 | 5
Period: Treatment Period , Switched to DE-111
Arm/Group | Allocated to Tafluprost | Allocated to Timolol | Allocated to Tafluprost + Timolol
Started | 48 | 45 | 43
Completed | 43 | 36 | 31
Not Completed | 5 | 9 | 12
Not completed — Adverse Event | 1 | 4 | 3
Not completed — Lack of Efficacy | 0 | 1 | 2
Not completed — Physician Decision | 0 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- DE-111: Switched to DE-111 ophthalmic solution (one drop at a time, once daily, bilateral topical instillation) from Tafluprost ophthalmic solution 0.0015% (one drop at a time, once daily, bilateral topical instillation), Timolol ophthalmic solution 0.5% (one drop at a time, BID, bilateral topical instillation), or concomitant Tafluprost ophthalmic solution 0.0015% plus Timolol ophthalmic solution 0.5% .
Arm/Group | DE-111
Number analyzed (Participants) | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 62
  >=65 years | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 55
Region of Enrollment [Number; unit: participants]
  Japan | 136

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in IOP (Intraocular Pressure) at End of Study
Time Frame: Treatment period: Week 0 (Baseline) and Week 52 (End of Study)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DE-111
Number analyzed (Participants) | 136
mmHg | -1.8 (2.2)

ADVERSE EVENTS:
Time Frame: Treatment period: Week 0 (Baseline) and Week 52 (End of Study)
Arm/Group | DE-111
Serious Adverse Events (participants affected / at risk) | 6/136
Other Adverse Events (participants affected / at risk) | 68/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DE-111 (N=136)
Acute myocardial infarction (Cardiac disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DE-111 (N=136)
Blepharal pigmentation (Eye disorders) | 9
Growth of eyelashes (Eye disorders) | 33
Punctate keratitis (Eye disorders) | 15
Conjunctival hyperaemia (Eye disorders) | 13
Nasopharyngitis (Eye disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No